CLINICAL TRIAL: NCT07200908
Title: A Global, Randomized, Open-label, Multicenter Phase 3 Trial Evaluating BJT-778 vs Bulevirtide for the Treatment of Chronic Hepatitis Delta Infection (AZURE-2)
Brief Title: A Trial Evaluating Brelovitug (BJT-778) vs Bulevirtide for the Treatment of Chronic Hepatitis Delta Infection (AZURE-2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bluejay Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJT-778-302; 2024-517167-23-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-16; First posted 2025-10-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepatitis D Infection
Keywords: Hepatitis Delta virus, HDV, Hepatitis D infection; Hepatitis D virus
MeSH Terms: conditions — Hepatitis D | interventions — bulevirtide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brelovitug (Experimental): Participants will receive treatment with brelovitug 300 mg once weekly for 96 weeks
  Interventions: Drug: Brelovitug 300 mg
- Bulevirtide for 48 weeks followed by brelovitug for 48 weeks (Active Comparator): Participants will receive bulevirtide 2 mg subcutaneously once daily for 48 weeks, followed by brelovitug 300 mg subcutaneously once weekly for the next 48 weeks.
  Interventions: Drug: Bulevirtide 2 mg and Brelovitug - 300 mg

INTERVENTIONS:
Drug: Brelovitug 300 mg — Route of administration- Subcutaneous Injection
  Other Names: BJT-778; BTG
  Arms: Brelovitug
Drug: Bulevirtide 2 mg and Brelovitug - 300 mg — Route of Administration- Subcutaneous Injection
  Other Names: Hepcludex
  Arms: Bulevirtide for 48 weeks followed by brelovitug for 48 weeks

SUMMARY:
This is a Phase 3, global, randomized, open-label, multicenter, trial evaluating brelovitug (BJT-778) vs bulevirtide for the treatment of chronic hepatitis delta infection (CHD). The main goal of this study is to test the effectiveness of brelovitug compared to bulevirtide as a long-term treatment in patients with chronic HDV infection.

DETAILED DESCRIPTION:
Study consists of 2 arms. Approximately 172 participants will be randomized 3:1 to one of the following treatment arms:

Arm 1: Participants will receive brelovitug 300 mg subcutaneously once weekly for 96 weeks.

Arm 2: Participants will receive bulevirtide 2 mg subcutaneously once daily for 48 weeks, followed by brelovitug 300 mg subcutaneously once weekly for the next 48 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Chronic HDV infection
3. HDV RNA >500 IU/mL at Screening
4. ALT >ULN at Screening
5. Willing to take or already taking HBV neucleos(t)ide therapy.

Key Exclusion Criteria:

1. Pregnant or nursing females
2. Unwilling to comply with contraception requirements during the study
3. Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy
4. Clinical hepatic decompensation (i.e., ascites, encephalopathy variceal hemorrhage).
5. Solid organ or bone marrow transplantation
6. Presence of other liver disease(s) (non-HBV/HDV), such as nonalcoholic steatohepatitis (NASH), alcohol associated hepatitis, cholestatic liver disease, hepatocellular carcinoma.

Note - Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with a composite endpoint of virologic response and ALT normalization | Week 48
  The composite endpoint is defined as virologic response (undetectable HDV RNA, < the lower limit of quantification [LLOQ], target not detected [TND]) and ALT normalization (decrease in ALT from baseline to ≤ upper limit of normal [ULN])

SECONDARY OUTCOMES:
Percentage of participants with treatment-emergent adverse events (TEAEs) | Up to 96 weeks
  An AE is any symptom, physical sign, syndrome, or disease that either emerges during the study or, if present at Screening (e.g., medical history), worsens during the study (post-Baseline/ Day 1), regardless of the suspected cause of the event.
Percentage of participants who discontinue treatment due to an adverse event (AE) | Up to 96 weeks
  An AE is any symptom, physical sign, syndrome, or disease that either emerges during the study or, if present at Screening (e.g., medical history), worsens during the study (post-Baseline/ Day 1), regardless of the suspected cause of the event.
Percentage of participants with HDV RNA ≥ 2 log10 IU/mL decline from baseline or TND | Up 96 Weeks
Percentage of participants with HDV RNA <LLOQ | Up to 96 Weeks
Percentage of participants with HDV RNA <LLOQ, TND | Up to 96 Weeks
Percentage of participants with ALT normalization | Up to 96 Weeks
  ALT normalization is defined as a decrease in ALT from baseline to ≤ ULN
Percentage of participants with ALT normalization in combination with virologic response of HDV RNA ≥ 2 log10 IU/mL decline from baseline or TND | Up to 96 Weeks
  The composite of participants with ALT normalization (decrease in ALT from baseline to ≤ ULN) and virologic response of HDV RNA ≥ 2 log10 IU/mL decline from baseline or TND.
Percentage of participants with ALT normalization in combination with HDV RNA <LLOQ | Up to 96 Weeks
  The composite of participants with ALT normalization (decrease in ALT from baseline to ≤ ULN) and virologic response of HDV RNA <LLOQ.
Percentage of participants with ALT normalization in combination with HDV RNA <LLOQ, TND | Up to 96 Weeks
  The composite of participants with ALT normalization (decrease in ALT from baseline to ≤ ULN) and virologic response of HDV RNA <LLOQ, TND.
Change from baseline in liver stiffness as determined by transient elastography (e.g., FibroScan) | Up to 96 Weeks
Change from baseline in APRI (AST-to-platelet ratio index) | Up to 96 Weeks
Change from baseline in CTP score in participants with cirrhosis | Up to 96 Weeks
Change from baseline in Model for End-Stage Liver Disease (MELD) score in participants with cirrhosis | Up to 96 Weeks
Percentage of participants with clinical disease progression from baseline in HDV-associated liver disease. | Up to 96 Weeks
  Liver disease progression will be determined by the Independent Data Monitoring Committee (IDMC).
Percentage of participants with HDV RNA <LLOQ, TND at post-treatment follow up. | Post-Treatment Weeks 24 and 48
Change from baseline in Health-Related Quality of Life (HRQoL) as measured by the Chronic Liver Disease Questionnaire-HBV (CLDQ-HBV) | Up to 96 Weeks
Change from baseline in Health-Related Quality of Life (HRQoL) as measured by the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | Up to 96 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bluejay Therapeutics, Study Director — Bluejay Therapeutics
Locations (20):
- Medical University of Graz, Graz, Austria
- Czechia (4):
  - Fakultni Nemocnice Brno, Brno, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové, Hradec Králové
  - Institute For Clinical And Experimental Medicine, Prague, Prague
  - Klin Med s.r.o., Prague, Prague
- Germany (2):
  - Goethe University Frankfurt, Frankfurt, Frankfurt
  - Rostock University Medical Center, Rostock, Rostock
- Romania (3):
  - National Institute Of Infectious Diseases, Bucharest, Bucharest
  - Spitalul Clinic De Boli Infectioase Si Tropicale Dr. Victor Babes, Bucharest, Bucharest
  - Centrul Medical Unirea S.R.L, Iași, Lasi
- Spain (2):
  - Hospital Universitario Torrecardenas, Almería, Almeria
  - Hospital Universitari Vall D Hebron, Barcelona, Barcelona
- Switzerland (2):
  - Hôpitaux Universitaires, Geneva, Canton of Geneva
  - HOCH Health Ostschweiz, Sankt Gallen, St.Gallen
- United Kingdom (6):
  - Queen Elizabeth Hospital Birmingham, Birmingham, Birmingham
  - Chelsea and Westminster Hospital NHS Foundation Trust, London, London
  - North Manchester General Hospital, Manchester, Manchester
  - Hull University Teaching Hospitals, Cottingham
  - Barts Health NHS Trust, London
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No